CLINICAL TRIAL: NCT00049088
Title: A Phase 1 Study of PS-341 in Combination With Docetaxel in Patients With Advanced Solid Tumors
Brief Title: Bortezomib and Docetaxel in Treating Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02508; J0203; U01CA070095 (NIH); CDR0000257807 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Docetaxel; Bevacizumab

ARMS (1):
- Treatment (docetaxel, bevacizumab) (Experimental): For course 1, patients receive docetaxel IV over 1 hour on days 1 and 8 and bortezomib IV over 3-5 seconds on days 9 and 12. Patients then receive 1 week of rest. For course 2 and all subsequent courses, patients receive docetaxel on days 1 and 8 and bortezomib on days 2, 5, 9, and 12. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 2-6 patients receive escalating doses of bortezomib and docetaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 1 of 6 patients experiences dose-limiting toxicity.
  Interventions: Drug: docetaxel; Biological: bevacizumab; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Phase I trial to study the effectiveness of combining bortezomib with docetaxel in treating patients who have advanced solid tumors. Bortezomib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining bortezomib with docetaxel may kill more tumor cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of bortezomib and docetaxel in patients with advanced solid tumors.

II. Determine the toxicity and tolerability of this regimen in these patients. III. Determine the biologic correlates of proteasome inhibition of bortezomib and determine the effects of this inhibition on the pharmacokinetics of docetaxel in these patients.

IV. Determine the antitumor efficacy of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

For course 1, patients receive docetaxel IV over 1 hour on days 1 and 8 and bortezomib IV over 3-5 seconds on days 9 and 12. Patients then receive 1 week of rest. For course 2 and all subsequent courses, patients receive docetaxel on days 1 and 8 and bortezomib on days 2, 5, 9, and 12. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 2-6 patients receive escalating doses of bortezomib and docetaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 1 of 6 patients experiences dose-limiting toxicity.

PROJECTED ACCRUAL: A minimum of 24 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor for which standard curative or palliative measures do not exist or are no longer effective

  * Metastatic or unresectable disease
* No known brain metastases
* Performance status - ECOG 0-2
* Performance status - Karnofsky 50-100%
* More than 12 weeks
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8 g/dL
* Bilirubin normal
* AST and ALT no greater than 1.5 times upper limit of normal (ULN) and alkaline phosphatase no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 5 times ULN (unless bone-derived) and AST and ALT less than 1.5 times ULN
* Creatinine normal
* Creatinine clearance at least 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study
* No prior allergic reactions attributed to taxanes (e.g., docetaxel or paclitaxel) or compounds of similar chemical or biological composition
* No prior allergic reactions to compounds similar to bortezomib or other study agents
* No known hypersensitivity to corticosteroids
* No predicted intolerance to regular, repeated administration of corticosteroids (e.g., poorly controlled diabetes or significant osteoporosis/osteopenia)
* No ongoing or active infection
* No other uncontrolled concurrent illness that would preclude study participation
* No psychiatric illness or social situation that would preclude study participation
* No peripheral neuropathy grade 2 or greater
* At least 4 weeks since prior chemotherapy (6 weeks for carmustine, nitrosoureas, or mitomycin) and recovered

  * No more than 3 courses of mitomycin
* Prior taxanes allowed

  * At least 6 months since prior docetaxel administered on a weekly schedule
* At least 4 weeks since prior radiotherapy and recovered
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer agents or therapies (commercial or investigational)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2002-08; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) based on the incidence of dose-limiting toxicity (DLT) as assessed by the NCI Common Toxicity Criteria (CTC) version 2.0 | 21 days
Toxicity and tolerability as assessed by NCI CTC version 2.0 | Up to 30 days after completion of study treatment

SECONDARY OUTCOMES:
Pharmacokinetics of docetaxel | At baseline, at 30 and 60 during infusion, at 10 min, 30 min, 1, 3, 7.5, 24, and 48 hours, and at 8 days after completion of docetaxel infusion
Response rate | Up to 30 days after completion of study treatment
20S proteasome activity | At 1 hour after first PS-341 infusion (week 2, day 2), and at 24 and 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Armstrong, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States